CLINICAL TRIAL: NCT03863275
Title: Analysis of Muscle Activity With Myofunctional Devices, Using Surface Electromyography
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fundación Universitaria CIEO (Other)
Responsible Party: Principal Investigator, Carolina Alvarez, Principal Investigator, Fundación Universitaria CIEO
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Electromyography
Record Dates: First submitted 2019-02-22; First posted 2019-03-05 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-02

CONDITIONS: Class II Malocclusion
MeSH Terms: conditions — Overbite | interventions — Observation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No intervation (Other): Children between the ages of 7 and 12 diagnosed with class II dental classification, who attend the Leonardo Da Vinci School after carrying out an intraoral and extraoral photography study and diagnostic impressions with study models accepting participation in the study, Children over the age of 12 who have an agreement according to the results of medical care. Patients with Pierre Robin syndrome or any form of cleft.
  Interventions: Other: Diagnosis and observation
- Myofunctional apparatus (Experimental): Boys and girls between 7 and 12 years skeletal class II, for the study group the individuals will be selected from the UNICIEO postgraduate clinic of orthopedic clinic orthodontics after conducting a full clinical case study exposed to a board of specialist teachers in orthodontics, where by means of several diagnostic methods a skeletal class II is confirmed that involves a treatment with myofunctional apparatus SN1; patients presenting syndromes that generate craniofacial alterations, patients with previous orthopedic treatment, patients with signs of condyle lesions, patients with Pierre Robin syndrome or any form of slit will be excluded.
  Interventions: Device: functional apparatus

INTERVENTIONS:
Device: functional apparatus — The EMG activity will be recorded during different shots: T0. The activity of the muscles of the mastication in the position of clinical rest for a minute, in maximum intercuspidation. (It will be measured with a dynamometer to standardize the force), and with the use of the equipment. T1 The patient's citation is scheduled six months after the use of myofunctional device Sn1 and the test will be performed again measuring electrical activity of right and left masseter and right and left temporal muscle at clinical rest for one minute, in maximum intercuspation, and with the use of the equipment To avoid the effects of fatigue, a rest period of at least 5 minutes between each of the recordings will be allowed
  Arms: Myofunctional apparatus
Other: Diagnosis and observation — Six months of observation in the control group: patients group the efforts are controlled. to obtain models and have an observation of the molar classification, and to verify if the terms of the inclusion in the study are taken into account, once it is confirmed that the activity is observed in the muscular activity of the chewing muscles, in two stages , at the beginning of the session and six months later. .
  Arms: No intervation

SUMMARY:
Importance and justification The importance of carrying out this study is to verify the electrical activity generated by the masticatory muscles to be able to have clarity of their performance in the development of orthopedic treatment, thus complementing the diagnosis to achieve a more successful treatment with myofunctional device SN1 in Class II malocclusions.

In addition, with the results of this study, treatment prediction criteria are provided to the clinician, depending on the thickness of the muscle, more specific equipment will be chosen to solve the malocclusion and prognosis when using the SN1 myofunctional device in class II malocclusions.

Additionally, it has academic utility, since there is little scientific evidence about myofunctional SN1 device and its impact on masticatory muscles, thus opening the door to a line of research where this study can be used as a basis for future orthopedic clinical research. in UNICIEO.

Added to this and according to the results, the knowledge about the SN1 will be updated, thus providing evidence for the teaching of orthopedics for the students; and also a measurement protocol with electromyography for children will be provided Overall objective To evaluate the electrical activity of the masseter and temporal muscles in patients from 7 to 12 years of age, with skeletal class II who are under treatment with myofunctional apparatus (Sn1), in the UNICIEO orthopedics clinic by means of kinesiological electromyography compare with a control group without use of the device Specific objectives

* Determine the activity of the masseter and temporal muscles of patients at rest (without functional orthopedic apparatus) in the two study groups.
* To determine the activity of the masseter and temporal muscles of the patients after the use of functional orthopedic equipment (Sn1), after six months of treatment and in the control group without treatment.

DETAILED DESCRIPTION:
Study design Prospective nonrandomized controlled clinical trial, 1: 1 allocation Participants Study group. Boys and girls between 7 and 12 years skeletal class II, for the study group the individuals will be selected from the UNICIEO postgraduate clinic of orthopedic clinic orthodontics after conducting a full clinical case study exposed to a board of specialist teachers in orthodontics, where by means of several diagnostic methods a skeletal class II is confirmed that involves a treatment with myofunctional apparatus SN1; patients presenting syndromes that generate craniofacial alterations, patients with previous orthopedic treatment, patients with signs of condyle lesions, patients with Pierre Robin syndrome or any form of slit will be excluded.

Control group. Children aged between 7 and 12 years diagnosed with class II dental classification, who attend the Leonardo Da Vinci School after carrying out an intraoral and extraoral photography study and diagnostic impressions with study models accepting participation in the study, children over the age of 12 will have to sign an agreement, patients who present syndromes that generate craniofacial alterations, patients with previous orthopedic treatment, patients with Pierre Robin syndrome or any form of slit will be excluded.

Interventions or independent variables

* Use of Sn1 equipment in the study group: the study participants are placed, which correspond to the study group, the Sn1 apparatus of which is composed of dorsal arches with an hourly intensity of 12 hours a day, where a control will be carried out monthly.
* Six months of observation in the control group: patients in the control group will be given informed consent, children over the age of 12 will have to sign an informed consent, then a photographic study of intraoral and extraoral photos will be made, impressions to obtain models and have an observation of the molar classification, and verify if it has the inclusion criteria of the study, once that participation is confirmed, the muscular activity of the masticatory muscles will be observed, in two times, at the beginning and at six months after.

Results or dependent variables.

Masseter and temporal muscle activity measured with EMG (microvolts) in the following moments:

Moment of measurement: the electrical activity will be taken at 2 moments of the study.

T0: Initial Moment

1. Rest: A record of electromyography will be taken where the patient has a natural position of the head and is in complete rest, resting time (60 seconds)
2. Maximum intercuspidation: The patient will be instructed to perform a force that will be measured with a dynamometer where it generates a dental tightening, to verify the electrical activity that is generated in that maximum contraction of masseter muscles captured by the electromyograph.
3. Use of the device: a record of the muscular activity will be made at the moment the patient puts on the Sn1 device.

T1: six months of use of functional equipment (Sn1)

1. Rest: A record of electromyography will be taken where the patient has a natural position of the head and is in complete rest, resting time (60 seconds)
2. Maximum intercuspidation: The patient will be instructed to perform a force that will be measured with a dynamometer where it generates a dental tightening, to verify the electrical activity that is generated in that maximum contraction of masseter muscles captured by the electromyograph.
3. Use of equipment (study group) will be a record of muscle activity at the time the patient puts on the Sn1 device

Sample size To date, no similar studies have been located, therefore a pilot test will be carried out with 10 patients from each group and with the result the sample size of the study will be calculated.

Statistical Methods The data will initially be tested using the Shapiro-Wilk test. Maximum changes in molar bite force during treatment or observation (T0 - T1) will be evaluated, and t-paired tests will be used to evaluate the statistical significance within each group. A comparison of the changes between the treatment and control groups will also be carried out using t-unpaired tests. Parametric analyzes will be used: Anova, Multivariate analysis of variance (Manova), T2 Hotelling test. All correlations were considered significant with p <0.05.

ELIGIBILITY:
Inclusion Criteria:

* Boys and girls from 7 to 12 years old with class II skeletal classification attending a consultation in the dental clinic of the UNICIEO foundation, to be fitted with myofunctional apparatus type Sn1

Exclusion Criteria:

* Patients who have had previous orthopedic treatment
* Patients with signs of condyle injuries
* Patients of Pierre Robin or any form of cleft
* Patients with syndromes that associate craniofacial anomalies and muscle alterations.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2019-02-26 (Estimated); Primary Completion 2019-08-26 (Estimated); Study Completion 2020-07-26 (Estimated)

PRIMARY OUTCOMES:
resting muscle activity, initial moment | 15 seconds
  Initial Moment . Measure with electromyography in microvolts
muscle activity in maximum intercuspidation, second moment | 10 seconds
  Measure with electromyography in microvolts.the maximum intercupidation is measured with a dynamometer
muscle activity with myofunctional apparatus, third moment | 10 seconds
  Measure with electromyography in microvolts.

CONTACTS AND LOCATIONS:
Overall Officials: carolina alvarez, dra, Principal Investigator — 35195385

IPD SHARING:
Plan to Share IPD: No